CLINICAL TRIAL: NCT02277639
Title: Phase I/II Study of Reduced Intensity Conditioning for Patients With Non-Malignant Diseases Using CD3+/CD19+ Depleted Unrelated Donor or Partially Matched Related Donor Peripheral Stem Cells
Brief Title: Reduced Intensity Conditioning Using CD3+/CD19+ Depletion for Non Malignant Transplantable Diseases
Acronym: MiniClini
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Nancy Bunin, BMT Medical Director, Children's Hospital of Philadelphia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-008330; CHP 980 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2014-10-22; First posted 2014-10-29 (Estimated); Results first posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-03

CONDITIONS: Bone Marrow Failure Syndromes; Immunodeficiencies; Immune Dysregulation Syndromes
Keywords: Transplant related mortality; Graft versus host disease; Bone marrow transplant
MeSH Terms: conditions — Bone Marrow Failure Disorders; Immunologic Deficiency Syndromes; Graft vs Host Disease

STUDY DESIGN:
Intervention Model Description: Reduced intensity conditioning with chemotherapy followed by stem cell transplant using the CliniMACs device to deplete CD3+ CD19+ peripheral stem cells.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bone Marrow Failure Syndrome (Experimental): Reduced intensity conditioning with chemotherapy followed by stem cell transplant using the CliniMACs device to deplete CD3+ CD19+ peripheral stem cells. Reduced intensity conditioning will include Busulfan, Fludarbine, Cyclophosphamide followed by stem cell infusion.
  Interventions: Device: CliniMACs device
- Immunodeficiency / Dysregulation (Experimental): Reduced intensity conditioning with chemotherapy followed by stem cell transplant using the CliniMACs device to deplete CD3+ CD19+ peripheral stem cells. Reduced intensity conditioning will include Busulfan, Fludarbine, Cyclophosphamide followed by stem cell infusion.
  Interventions: Device: CliniMACs device

INTERVENTIONS:
Device: CliniMACs device — Reduced intensity conditioning with chemotherapy followed by stem cell transplant using the CliniMACs device to deplete CD3+ CD19+ peripheral stem cells.

SUMMARY:
This is a Phase II trial to determine the ability of a reduced intensity conditioning regimen to allow successful engraftment with CD3+ /CD19+ depleted peripheral stem cell grafts from mismatched donors. There are two conditioning regimens depending upon patient diagnosis and age.

DETAILED DESCRIPTION:
This study will allow transplantation using a reduced intensity conditioning regimen for children with non-malignant diseases who lack a matched related or unrelated donor. Donors will be unrelated or partially matched related, depending upon urgency and availability. If each parent is haploidentical, the mother will be preferred, as there is evidence of reduced transplant related mortality and superior survival with a maternal donor. The risks of severe graft vs host disease (GVHD) and Epstein-Barr lymphoproliferative disorder will be reduced or eliminated by T and B cell depletion using the Miltenyi Clinimacs device. Patients with bone marrow failure syndromes, who are at high risk for rejection, will undergo pre-conditioning immune suppression with Thymoglobulin. It is recommended that patients with immunedysregulation syndromes receive pre-RIC alemtuzumab as this may reduce the risk on non-engraftment and hyperinflammatory states.

Post-transplant immune suppression will be used to prevent GVHD, as CD3 depletion does not deplete as completely as CD34+ selection. It will be rapidly weaned if no GVHD by day 100 to allow immune reconstitution.

ELIGIBILITY:
Inclusion Criteria:

* Bone marrow failure syndromes for which SCT is indicated, including severe aplastic anemia refractory to non transplant therapies congenital neutropenia, congenital thrombocytopenia, congenital red cell aplasia
* Immunodeficiencies for which allogeneic hematopoietic stem cell transplant is indicated, including severe combined immunodeficiencies, Wiskott-Aldrich syndrome, IPEX syndrome, X-linked lymphoproliferative disease
* Immune dysregulation syndromes, including refractory or recurrent hemophagocytic lymphohistiocytosis, HLH with genetic mutations, refractory multisystemic Langerhans cell histiocytosis, other MAS refractory to standard therapy
* Organ function clearance

Exclusion Criteria:

* Uncontrolled bacterial, viral or fungal infections
* HLA matched related or unrelated donor able to donate mobilized peripheral stem cells.
* Fanconi's syndrome, dyskeratosis congenita or other chromosomal fragility syndromes
* Pregnant Females

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2011-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Bunin, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bone Marrow Failure Syndrome; Immunodeficiency / Dysregulation: Reduced intensity conditioning with chemotherapy followed by stem cell transplant using the CliniMACs device to deplete CD3+ CD19+ peripheral stem cells. Reduced intensity conditioning will include Busulfan, Fludarbine, Cyclophosphamide followed by stem cell infusion.
  CD3+/CD19+ delpletion using CliniMACs device follwing reduced intensity conditioning: Reduced intensity conditioning with chemotherapy followed by stem cell transplant using the CliniMACs device to deplete CD3+ CD19+ peripheral stem cells.
Period: Overall Study
Arm/Group | Bone Marrow Failure Syndrome | Immunodeficiency / Dysregulation
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bone Marrow Failure Syndrome | Immunodeficiency / Dysregulation | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Continuous [Median (Full Range); unit: years] |  | 9.5 [4 to 15] | 9.5 [4 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Engraftment
Description: The primary objective is to determine event free survival with durable stable engraftment of donor cells at one year.
Time Frame: One Year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Failure Syndrome | Immunodeficiency / Dysregulation
Number analyzed (Participants) | 0 | 2
Participants |  | 2

ADVERSE EVENTS:
Arm/Group | Bone Marrow Failure Syndrome | Immunodeficiency / Dysregulation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No